CLINICAL TRIAL: NCT01898442
Title: Pharmacodynamic Profiles of Ticagrelor in Patients With ST Elevation Myocardial Infarction: A Randomized Comparison of Different Loading Dosage Regimens
Brief Title: High Ticagrelor Loading Dose in STEMI
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: University of Florida (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: TicagSTEMI
Record Dates: First submitted 2013-07-01; First posted 2013-07-12 (Estimated); Results first posted 2015-06-08 (Estimated); Last update posted 2015-06-08 (Estimated); Status verified 2014-06

CONDITIONS: Coronary Artery Disease
Keywords: platelet function; ticagrelor; STEMI
MeSH Terms: conditions — Coronary Artery Disease; ST Elevation Myocardial Infarction | interventions — Ticagrelor

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: Yes

ARMS (3):
- Ticagrelor 180 (Active Comparator): Standard ticagrelor 180mg loading dose
  Interventions: Drug: Ticagrelor 180mg
- Ticagrelor 270mg (Experimental): High ticagrelor 270mg loading dose
  Interventions: Drug: Ticagrelor 270mg
- Ticagrelor 360mg (Experimental): High ticagrelor 360mg loading dose
  Interventions: Drug: Ticagrelor 360mg

INTERVENTIONS:
Drug: Ticagrelor 180mg — Rndomization to standard or high ticagrelor loading dose regimens
  Other Names: Brilinta
  Arms: Ticagrelor 180
Drug: Ticagrelor 270mg — Randomization to standard or high loading dose regimen
  Other Names: Brilinta
  Arms: Ticagrelor 270mg
Drug: Ticagrelor 360mg — Randomization to standrad or high loading dose regimen
  Other Names: Brilinta
  Arms: Ticagrelor 360mg

SUMMARY:
Ticagrelor is a reversible direct acting P2Y12 antagonist, which has shown to be superior to clopidogrel, in adjunct to aspirin, in preventing recurrent ischemic events. Ticagrelor is considered a first line therapy to be administered as soon as possible in ACS patients. However, the pharmacodynamic effects of ticagrelor at the recommended 180mg loading dose are delayed in patients with STEMI undergoing primary PCI. The use of higher loading dose regimens of ticagrelor has therefore been advocated. The proposed investigation will have a prospective, randomized, parallel design in which STEMI patients undergoing primary PCI will be randomized to receive three different loading dose of ticagrelor (180 mg, 270 mg and 360 mg). Pharmacodynamic testing will be performed at several time points to test our study hypothesis that a higher loading dose regiment will achieve more promptly enhanced platelet inhibitory effects.

DETAILED DESCRIPTION:
Dual antiplatelet therapy consisting of aspirin and a P2Y12 receptor antagonist is the cornerstone of treatment for prevention of thrombotic events in patients with acute coronary syndromes (ACS). Ticagrelor is a reversible direct acting P2Y12 antagonist, which has shown to be superior to clopidogrel, in adjunct to aspirin, in preventing recurrent ischemic events, including cardiovascular mortality. Ticagrelor was recently approved for clinical use in ACS patients, at a dose of 180 mg loading dose and 90 mg twice/day maintenance dose. Ticagrelor is considered a first line therapy to be administered as soon as possible in ACS patients, including those presenting with ST-elevation myocardial infarction (STEMI) undergoing primary percutaneous coronary intervention (PCI). However, there are discordant data on the onset of its antiplatelet effects in this particular setting. In particular, the pharmacodynamic effects of ticagrelor at the recommended 180mg loading dose are delayed in patients with STEMI undergoing primary PCI. The use of higher loading dose regimens of ticagrelor has therefore been advocated. However, if the administration of a higher ticagrelor loading dose may overcome this limitation is still unknown and represents the aim of our study. The proposed investigation will have a prospective, randomized, parallel design in which STEMI patients undergoing primary PCI will be randomized to receive three different loading dose of ticagrelor (180 mg, 270 mg and 360 mg). Pharmacodynamic testing will be performed at several time points to test our study hypothesis that a higher loading dose regiment will achieve more promptly enhanced platelet inhibitory effects. This study will provide insights on the pharmacodynamic effects of higher ticagrelor loading doses and will help clinicians choose the most appropriate treatment to avoid complications related to inadequate platelet inhibition in the early phase of patients with STEMI undergoing primary PCI.

ELIGIBILITY:
Inclusion Criteria:

* Patients with ST-elevation myocardial infarction undergoing primary PCI.
* Age between 18 and 80 years old.

Exclusion Criteria:

* History of prior intracranial bleeding.
* On treatment with a P2Y12 receptor antagonist (ticlopidine, clopidogrel, prasugrel, ticagrelor) in past 30 days.
* Known allergies to aspirin or ticagrelor.
* On treatment with oral anticoagulant (Vitamin K antagonists, dabigatran, rivaroxaban).
* Treatment with IIb/IIIa glycoprotein inhibitors.
* Fibrinolytics within 24 hours
* Known blood dyscrasia or bleeding diathesis.
* Known platelet count <80x106/mL.
* Known hemoglobin <10 g/dL.
* Active bleeding.
* Hemodynamic instability.
* Known creatinine clearance <30 mL/minute.
* Known severe hepatic dysfunction.
* Patients with sick sinus syndrome (SSS) or high degree AV block without pacemaker protection.
* Current treatment with drugs interfering with CYP3A4 metabolism (to avoid interaction with Ticagrelor): Ketoconazole, itraconazole, voriconazole, clarithromycin, nefazodone, ritonavir, saquinavir, nelfinavir, indinavir, atazanavir, and telithromizycin.
* Pregnant females*.

  * Women of childbearing age must use reliable birth control (i.e. oral contraceptives) while participating in the study.

Ages: 18 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 52 (Actual)
Dates: Start 2013-09; Primary Completion 2014-06 (Actual); Study Completion 2014-06 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Dominick Angiolillo, MD, PhD, Principal Investigator — University of Florida
Locations (1):
- University of Florida, Jacksonville, Florida, United States

REFERENCES:
- [Derived] Franchi F, Rollini F, Cho JR, Bhatti M, DeGroat C, Ferrante E, Dunn EC, Nanavati A, Carraway E, Suryadevara S, Zenni MM, Guzman LA, Bass TA, Angiolillo DJ. Impact of Escalating Loading Dose Regimens of Ticagrelor in Patients With ST-Segment Elevation Myocardial Infarction Undergoing Primary Percutaneous Coronary Intervention: Results of a Prospective Randomized Pharmacokinetic and Pharmacodynamic Investigation. JACC Cardiovasc Interv. 2015 Sep;8(11):1457-1467. doi: 10.1016/j.jcin.2015.02.030. PMID 26404199

RESULTS

PARTICIPANT FLOW:
Recruitment Details: Between September 2013 and June 2014.
Pre-assignment Details: There were a total of 129 STEMI activations; of these, 52 patients provided their written informed consent to participate in the study and were randomized.
Groups:
- Ticagrelor 180mg: Standard ticagrelor 180mg loading dose
  Ticagrelor 180mg: Randomization to standard ticagrelor loading dose
- Ticagrelor 270mg: High ticagrelor 270mg loading dose
  Ticagrelor 270mg: Randomization to a high ticagrelor loading dose regimen
- Ticagrelor 360mg: High ticagrelor 360mg loading dose
  Ticagrelor 360mg: Randomization to a high ticagrelor loading dose regimen
Period: Overall Study
Arm/Group | Ticagrelor 180mg | Ticagrelor 270mg | Ticagrelor 360mg
Started | 17 | 17 | 18
Completed | 16 | 15 | 15
Not Completed | 1 | 2 | 3
Not completed — Hemolysis/technical problems | 1 | 2 | 2
Not completed — Patient vomited pills | 0 | 0 | 1

BASELINE CHARACTERISTICS:
Population: The primary population was used for analysis of baseline characteristics and primary and secondary endpoints. The primary population was defined as patients who received the randomized loading dose of study medication and had at least 75% of valid data, which needed to include the primary endpoint time point.
Groups:
- Total: Total of all reporting groups
Arm/Group | Ticagrelor 180mg | Ticagrelor 270mg | Ticagrelor 360mg | Total
Number analyzed (Participants) | 16 | 15 | 15 | 46
Age, Continuous [Mean (Standard Deviation); unit: years] | 60 (8.6) | 58 (8.5) | 57 (12.1) | 58 (9.5)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 2 | 5 | 7 | 14
  Male | 14 | 10 | 8 | 32
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0 | 0 | 0 | 0
  Asian | 0 | 0 | 0 | 0
  Native Hawaiian or Other Pacific Islander | 0 | 0 | 0 | 0
  Black or African American | 5 | 3 | 4 | 12
  White | 11 | 12 | 11 | 34
  More than one race | 0 | 0 | 0 | 0
  Unknown or Not Reported | 0 | 0 | 0 | 0

OUTCOME MEASURES:

1. Primary Outcome: Platelet Reactivity by VerifyNow P2Y12
Description: The primary end-point of the study was the comparison of the P2Y12 reaction units (PRU) determined by VerifyNow P2Y12 at 1 hour after administration
Time Frame: 1 hour
Measure: Least Squares Mean (Standard Error); unit: PRU
Arm/Group | Ticagrelor 180mg | Ticagrelor 270mg | Ticagrelor 360mg
Number analyzed (Participants) | 16 | 15 | 15
PRU | 188 (20) | 125 (23) | 228 (23)
Statistical Analysis 1: Comparison: Ticagrelor 180mg vs Ticagrelor 270mg vs Ticagrelor 360mg; Test type: Superiority or Other; p = 0.017, ANCOVA

2. Secondary Outcome: Platelet Reactivity by VerifyNow P2Y12 at Other Time Points
Description: Secondary outcomes included the comparison of the P2Y12 reaction units (PRU) determined by VerifyNow P2Y12 at 30 min and 2, 4, 8, 24 hours after ticagrelor loading dose administration
Time Frame: 30 min and 2, 4, 8, 24 hours
Measure: Least Squares Mean (Standard Error); unit: PRU
Arm/Group | Ticagrelor 180mg | Ticagrelor 270mg | Ticagrelor 360mg
Number analyzed (Participants) | 16 | 15 | 15
PRU
  30 min | 231 (15) | 225 (17) | 249 (17)
  2 hours | 90 (28) | 83 (31) | 148 (31)
  4 hours | 75 (19) | 46 (22) | 69 (22)
  8 hours | 60 (18) | 44 (21) | 78 (21)
  24 hours | 39 (13) | 41 (14) | 72 (14)

3. Secondary Outcome: Platelet Reactivity by Vasodilator-stimulated Phosphoprotein (VASP) at All Time Points
Description: Secondary outcomes included the comparison of the platelet reactivity index (PRI) determined by vasodilator-stimulated phosphoprotein (VASP) at 30 min and 1, 2, 4, 8, 24 hours after ticagrelor loading dose administration
Time Frame: 30 min and 1, 2, 4, 8, 24 hours
Measure: Least Squares Mean (Standard Error); unit: PRI
Arm/Group | Ticagrelor 180mg | Ticagrelor 270mg | Ticagrelor 360mg
Number analyzed (Participants) | 16 | 15 | 15
PRI
  30 min | 76 (6) | 81 (6) | 78 (6)
  1 hour | 56 (7) | 51 (8) | 78 (8)
  2 hours | 41 (9) | 39 (10) | 48 (10)
  4 hours | 35 (6) | 30 (7) | 21 (7)
  8 hours | 25 (5) | 30 (5) | 23 (5)
  24 hours | 27 (4) | 30 (5) | 28 (5)

4. Secondary Outcome: Pharmacokinetic Profiles of Ticagrelor (Tmax)
Description: Pharmacokinetic assessments included determination of plasma concentration of ticagrelor. Time for the maximum plasma concentration (Tmax), maximum observed plasma concentration (Cmax) and the area under the plasma concentration vs. time curve from time 0 to the last measurable concentration (AUC0-t) were calculated.
Time Frame: 24 hours
Measure: Geometric Mean (Full Range); unit: hours
Arm/Group | Ticagrelor 180mg | Ticagrelor 270mg | Ticagrelor 360mg
Number analyzed (Participants) | 16 | 15 | 15
hours | 3.9 [2 to 24] | 5.0 [1 to 24] | 7.4 [2 to 24]

5. Secondary Outcome: Pharmacokinetic Profiles of Ticagrelor (Cmax)
Description: as for outcome 4
Time Frame: 24 hours
Measure: Geometric Mean (Full Range); unit: ng/mL
Arm/Group | Ticagrelor 180mg | Ticagrelor 270mg | Ticagrelor 360mg
Number analyzed (Participants) | 16 | 15 | 15
ng/mL | 789 [95 to 3550] | 1208 [276 to 2940] | 1208 [242 to 4040]

6. Secondary Outcome: Pharmacokinetic Profiles of Ticagrelor (AUC0-t)
Description: as for outcome 4
Time Frame: 24 hours
Measure: Geometric Mean (Full Range); unit: ng*hr/mL
Arm/Group | Ticagrelor 180mg | Ticagrelor 270mg | Ticagrelor 360mg
Number analyzed (Participants) | 16 | 15 | 15
ng*hr/mL | 7893 [1270 to 33974] | 12379 [2935 to 33105] | 12381 [768 to 66201]

ADVERSE EVENTS:
Time Frame: In-hospital adverse events, including ischemic events, bleeding, bradyarrhythmias, and dyspnea, defined according to previously reported criteria in the PLATO trial, were recorded.
Arm/Group | Ticagrelor 180mg | Ticagrelor 270mg | Ticagrelor 360mg
Serious Adverse Events (participants affected / at risk) | 0/17 | 1/17 | 1/18
Other Adverse Events (participants affected / at risk) | 2/17 | 1/17 | 0/18
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Ticagrelor 180mg (N=17) | Ticagrelor 270mg (N=17) | Ticagrelor 360mg (N=18)
Ischemic stroke (Vascular disorders) | 0 (0) | 1 (1) | 0 (0) — One patients in the 270mg group developed a peri-PCI ischemic stroke, which was manged according to standard-of-care.
Major-life threatening bleed (Vascular disorders) | 0 (0) | 0 (0) | 1 (1) — One patient in the 360mg group experienced a major-life threatening bleed (hypovolemic shock requiring vasopressor and transfusion)
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Ticagrelor 180mg (N=17) | Ticagrelor 270mg (N=17) | Ticagrelor 360mg (N=18)
Minimal/minor bleeding (Vascular disorders) | 2 (2) | 1 (1) | 0 (0) — Vascular access-related bleeding

LIMITATIONS AND CAVEATS:
The study was not powered to assess safety or efficacy, which would require larger clinical studies. Although laboratory personnel were blinded to treatment assignment, the study had an open-label design.

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes